CLINICAL TRIAL: NCT00806559
Title: SIT Trial: The Effect of Clinical Room Design on the Quality of the Clinical Encounter
Brief Title: Space and Interaction Trial: Room Design and Patient-physician Interaction
Acronym: SIT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mayo Clinic (Other)
Collaborators: Steelcase (Industry)
Responsible Party: Victor Montori, M.D., Mayo Clinic
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Health Services Research
Other Study IDs: 07-000135
Record Dates: First submitted 2008-12-10; First posted 2008-12-11 (Estimated); Last update posted 2011-12-14 (Estimated); Status verified 2011-12

CONDITIONS: Internal Medicine Patients; Participating Staff
Keywords: effects clinical space; follow-up appointments

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Usual room (Active Comparator): Patients in this arm will see their clinician in the usual clinical exam room
  Interventions: Other: Control room
- Re-designed room (Experimental): Patients assigned to this arm will see the physician in a redesigned clinical exam room
  Interventions: Other: Re-designed room

INTERVENTIONS:
Other: Re-designed room — In the redesigned room patients and clinicians are sitting at a single table in a different configuration compared to the usual clinical exam room, with the doctor at the computer and two chairs for the patient and family/friends.
  Arms: Re-designed room
Other: Control room — This is the usual clinical room for a clinical visit, with physician at desk and chairs along the wall for patient/family.
  Arms: Usual room

SUMMARY:
The purpose of this study is to improve the clinical encounter through the design of the clinical environment. We will conduct a randomized controlled trial to measure the extent to which a newly designed clinical room, compared to a traditional room, affects the patient-physician interaction. We will judge this outcome by (a) videotaping encounters; and (b) conducting post-visit surveys with patients and an interview with physicians. We will use both qualitative and quantitative tools, including a validated and widely used interaction coding system on the videotapes, to draw inferences from these data.

ELIGIBILITY:
Eligible Clinicians:

1. In the Department of GIM or Preventive Medicine
2. Able and Willing to participate in research study.

Eligible patients:

1. Patient of a clinician participating in the study
2. 18 years or older
3. Seeing clinician for return/summary visit.

Exclusion Criteria:

1.) Not able to give informed consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2007-07; Primary Completion 2008-04 (Actual); Study Completion 2008-04 (Actual)

PRIMARY OUTCOMES:
Patient and Clinician Interaction variables (duration of the encounter, patient sense of control in encounter, patient's ability to access information from the computer monitor and the quality of the verbal and non-verbal interaction). | Immediately post clinical visit (survey)
Patient experience of the clinical encounter. The following variables will be measured: patient satisfaction with the room, patient satisfaction with the encounter and the quality of the relationship. | Immediately post visit

CONTACTS AND LOCATIONS:
Overall Officials: Victor M. Montori, M.D., MSc, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic, Rochester, Minnesota, United States

REFERENCES:
- [Derived] Almquist JR, Kelly C, Bromberg J, Bryant SC, Christianson TH, Montori VM. Consultation room design and the clinical encounter: the space and interaction randomized trial. HERD. 2009 Fall;3(1):41-78. doi: 10.1177/193758670900300106. PMID 21165880